CLINICAL TRIAL: NCT03504215
Title: Exercise Intervention to Rescue the Adverse Effect of Preterm Birth on Cardiovascular and Pulmonary Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Western University, Canada (Other); Université de Montréal (Other); Ottawa Hospital Research Institute (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Anne Monique NUYT,MD, Chief of Neonatalogy and Professor of Pediatrics, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HAPI Fit Clinical Study
Record Dates: First submitted 2018-04-10; First posted 2018-04-20 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Prematurity; Extreme
Keywords: extremely preterm; young adults; term; exercise capacity; pulmonary function; muscle oxygenation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Group assignments. Both groups are evaluated before and after a 14 week supervised exercise (aerobic and resistance training) intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- young adults (Experimental): Both young adults born preterm (n=60) and term (n=30) will undergo the exercise intervention.
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — Assigned intervention : 14-week supervised intervention of aerobic and resistance training.

SUMMARY:
In spite of advances in neonatal intensive care allowing the first generation survivors of extreme prematurity to now reach young adulthood, these individuals present with reduced exercise capacity; a strong predictor of later chronic disease and mortality. The reason why individuals born preterm have exercise limitation remains unclear and may be a consequence of impact of preterm birth and associated neonatal difficulties on the development of organs important for exercise, namely the lungs, the heart, the vessels (which bring blood and oxygen to the muscles) and the muscles. It is well known that exercise benefits overall health in at-risk as well diseased populations. However, whether exercise training can improve fitness in young adults born preterm was not demonstrated and whether the cardiovascular, pulmonary and muscle impairments associated with preterm birth are reversible through exercise intervention in young adulthood is unknown.

DETAILED DESCRIPTION:
The investigators postulate that a 14-week exercise intervention will improve exercise capacity in preterm adults, as seen in other at-risk populations, in correlation with measures of vascular health, heart and muscle perfusion and oxygenation, and pulmonary function detected by cutting edge and highly sensitive imaging and circulating biomarkers. These markers are more sensitive to pre-disease changes than traditional health measures, and are largely unexplored in preterm populations.

The investigators will:

1. Determine whether a 14-week supervised exercise training improves exercise capacity in young adults (18-29 years old) born very preterm at <29 weeks gestational age.
2. Examine whether improvement in exercise capacity is associated with changes in (a) markers of vascular health including circulating endothelial progenitor cells and microparticles, (b) cardiac perfusion by cutting-edge oxygenation-sensitive cardiovascular magnetic resonance imaging (MRI), (c) lung regional ventilation measured by newly developed hydrogen proton (1H) MRI, (d) muscle oxygenation during exercise.
3. Compare the response of the above measures to exercise intervention between young adults born very preterm and term controls.

ELIGIBILITY:
Inclusion Criteria:

Both groups :

* Aged between 18-29 years old
* Less than 120 minutes of exercise per week
* Willingness to be part of the 14 weeks exercise intervention

Preterm group:

- Born under 29 weeks of gestation

Term group :

* Born between 37-41 weeks
* Appropriate weight fo gestational weight

Exclusion Criteria:

* Pregnancy
* conditions excludins individual from exercise

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Measurement of the peak oxygen consumption before and after the physical intervention | 16 weeks
  Respiratory exchange ratio (RER) (%)
Measurement of the peak oxygen consumption before and after the physical intervention | 16 weeks
  Oxygen uptake (VO2max) (mL/min)
Measurement of the peak oxygen consumption before and after the physical intervention | 16 weeks
  Carbon dioxide production (VCO2) (L/min)
Measurement of the peak oxygen consumption before and after the physical intervention | 16 weeks
  VO2peak (mL/kg/min)
Measurement of the peak oxygen consumption before and after the physical intervention | 16 weeks
  Weight (kg)
Measurement of the peak oxygen consumption before and after the physical intervention | 16 weeks
  Height (cm)
Measurement of the peak oxygen consumption before and after the physical intervention | 16 weeks
  Age (years)

SECONDARY OUTCOMES:
Cardiac oxygen sensitive MRI (OS-MRI) | 18 weeks
  myocardial perfusion in response to CO2 modulation
Lung regional ventilation using a 3D proton MRI ultrashort ecotime | 1 week
  Parenchyma signal intensity (SI)
Muscle oxygenation | 18 weeks
  Near-infrared spectroscopy (NIRS)
Pulmonary function | 18 weeks
  Forced spirometry (FEV1, L)
Pulmonary function | 18 weeks
  Forced spirometry (FVC, L)
Pulmonary function | 18 weeks
  Forced spirometry (FEF25-75, L/s)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Monique Nuyt, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- St. Justine's Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Tardif CB, Mathieu ME, Caru M, Al-Simaani A, Girard-Bock C, Cloutier A, Stickland MK, Nuyt AM, Luu TM. HAPI Fit: An Exercise Intervention to Improve Peak Aerobic Capacity in Young Adults Born Very Preterm. Med Sci Sports Exerc. 2024 Jan 1;56(1):44-52. doi: 10.1249/MSS.0000000000003279. Epub 2023 Aug 30. PMID 37707478